CLINICAL TRIAL: NCT05374902
Title: Efficacy of Procedural Information, Buzzy, and Multiple Interventions on Pain Management in Undergoing Venipuncture Children: A Randomised Controlled Trial
Brief Title: Efficacy of Animation, Buzzy, and Multiple Interventions on Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Buket MERAL, Research Asistant, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BMERAL
Record Dates: First submitted 2022-04-19; First posted 2022-05-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Pain, Procedural; Child; Phlebotomy; Venipuncture
Keywords: procedural pain; child; phlebotomy; venipunctur; animation; nursing practice; Non-pharmacological method
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Masking Description: Single (investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Procedural informational animation group (Experimental): Children and parents have watched procedural informational animation before venipuncture. Afterward, the children and their parents entered the blood drawn unit, and the procedure was performed as in standard care.
  Interventions: Other: Providing procedural informational animation video
- Buzzy group (Experimental): Buzzy® was placed on the injection site and cold application and vibration were turned on 60 s before the procedure. Then, the nurse moved Buzzy® about 3-5 cm above the injection site. The procedure was performed with buzzy®. The Buzzy® intervention and phlebotomy were terminated at the same time.
  Interventions: Device: Buzzy
- Multiple interventions group (Experimental): Children and parents have watched procedural informational animation before venipuncture. Afterward, the children and their parents entered the blood drawn unit. Buzzy® was placed on the injection site and cold application and vibration were turned on 60 s before the procedure. Then, the nurse moved Buzzy® about 3-5 cm above the injection site. The procedure was performed with buzzy®. The Buzzy® intervention and phlebotomy were terminated at the same time.
  Interventions: Combination Product: Multiple interventions
- Control group (No Intervention): Children in this group received standard care. A local anesthetic is not used, and the parents are with their children during the procedure in the standard care of the blood collection unit

INTERVENTIONS:
Other: Providing procedural informational animation video — Children and parents have watched procedural informational animation before venipuncture. Afterward, the children and their parents entered the blood drawn unit, and the procedure was performed as in standard care.
  Arms: Procedural informational animation group
Device: Buzzy — Buzzy® was placed on the injection site and it was turned on 60 s before the procedure. Then, the nurse moved Buzzy® about 3-5 cm above the injection site. The procedure was performed with buzzy®. The Buzzy® intervention and phlebotomy were terminated at the same time.
  Arms: Buzzy group
Combination Product: Multiple interventions — Watching procedural informational animation video prior to venipuncture, and Buzzy application during venipuncture
  Arms: Multiple interventions group

SUMMARY:
The aim of the study was to determine the effects of providing procedural informational animation, Buzzy application during the procedure, the combination of both interventions (Animated video and Buzzy), and standard care on pain management during venipuncture in children aged 6-12 years.

DETAILED DESCRIPTION:
A prospective randomized controlled trial design was used to determine the effects of Buzzy, procedural informational animation, multiple interventions (Buzzy and Animated video), and standard care on the pain level of 6-12 years aged children during venıpunctrue. The study was conducted in the territory hospital pediatric blood collection unit The sample size was determined by power analysis and 45 child-parent pairs were included in each group. The patients who met the sample selection criteria were randomly and equally assigned into 4 groups using a computer-based program. As a data collection tools, Data Collection Form and Wong-Baker have been used. Venipuncture-related pain was self-reported by each child, as well as through parents and nurse. Children in the multiple interventions group were shown procedural informative animation and the venipunctıre procedure was performed with buzzy®. Standard care was applied to the control group, in which no local anesthetic was used and families could accompany the bloodletting process. The pain responses of the children were evaluated twice, immediately after the procedure (while the child was sitting in the blood collection chair) and 2-3 minutes after the procedure, both by the children's self-reports and by the parents and the nurse.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 6 and 12 years,
* admitted to the hospital as an outpatient,
* having complete skin integrity at the place where the Buzzy device will be inserted
* having the ability to verbally communicate
* parents being literate.

Exclusion Criteria:

* having any acute pain at the time of the procedure
* having any audiovisual, cognitive sensitivity, or physical disability and having a chronic or life-threatening disease
* being under the influence of any sedative/anticonvulsant/analgesic drug,
* getting blood drawn in the last month
* failure to phlebotomy at the first attempt
* having nerve damage or peripheral neuropathy.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Pain assessment | The pain was measured at 30 seconds after (immediately) the venipuncture.
  Pain intensity was assessed Wong-Baker FACES Pain Rating Scale. It is used to determine the pain level of children aged between 3 and 18 years through their facial expressions which are assigned the values of 0 and 10. The first face represents a pain score of 0, and indicates "no hurt". The last face represents a pain score of 10, and indicates "hurts worst."
Pain assessment | The pain was measured at 2-3 minutes after the venipuncture.
  Pain intensity was assessed Wong-Baker FACES Pain Rating Scale. It is used to determine the pain level of children aged between 3 and 18 years through their facial expressions which are assigned the values of 0 and 10. The first face represents a pain score of 0, and indicates "no hurt". The last face represents a pain score of 10, and indicates "hurts worst."

SECONDARY OUTCOMES:
Pain assessment - parent | The pain was measured at 30 seconds after (immediately) the venipuncture by parent
  Pain intensity was assessed Wong-Baker FACES Pain Rating Scale. It is used to determine the pain level of children aged between 3 and 18 years through their facial expressions which are assigned the values of 0 and 10. The first face represents a pain score of 0, and indicates "no hurt". The last face represents a pain score of 10, and indicates "hurts worst."
Pain assessment - parent | The pain was measured at 2-3 minutes after the venipuncture by parent
  Pain intensity was assessed Wong-Baker FACES Pain Rating Scale. It is used to determine the pain level of children aged between 3 and 18 years through their facial expressions which are assigned the values of 0 and 10. The first face represents a pain score of 0, and indicates "no hurt". The last face represents a pain score of 10, and indicates "hurts worst."
Pain assessment - nurse | The pain was measured at 30 seconds after (immediately) the venipuncture by nurse.
  Pain intensity was assessed Wong-Baker FACES Pain Rating Scale. It is used to determine the pain level of children aged between 3 and 18 years through their facial expressions which are assigned the values of 0 and 10. The first face represents a pain score of 0, and indicates "no hurt". The last face represents a pain score of 10, and indicates "hurts worst."
Pain assessment - nurse | The pain was measured at 2-3 minutes after the venipuncture by nurse.
  Pain intensity was assessed Wong-Baker FACES Pain Rating Scale. It is used to determine the pain level of children aged between 3 and 18 years through their facial expressions which are assigned the values of 0 and 10. The first face represents a pain score of 0, and indicates "no hurt". The last face represents a pain score of 10, and indicates "hurts worst."

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Bayburt University/Faculty of Health Sciences, Bayburt
  - Ordu University/Faculty of Medicine, Ordu
  - Karadeniz Technical University, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.